CLINICAL TRIAL: NCT00767702
Title: Exploring the Use of Population Descriptors in Human Genetic Research
Brief Title: Use of Population Descriptors in Human Genetic Research
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908217; 08-HG-N217
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2012-08-08

CONDITIONS: Population Groups; Genetics, Medical; Ethnology; Disease; Qualitative Research
Keywords: Genetic/Genomic Researchers; Human Genetic Variation; Interviews; Research Design; Race/Ethnicity; Interview
MeSH Terms: conditions — Disease

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will explore scientists opinions and practices regarding the use of population descriptors (e.g., race, ethnicity, ancestry, geography and nationality) to describe a research study population. It will collect genetic researchers opinions, understandings and experiences studying human genetics and genetic variation.

Scientists who are a principal investigator or co-principal investigator n a human genetic or genomic study of a common disease with at least preliminary data that uses population descriptors may be eligible for the study.

Participants are asked to think about their study populations and how they are described in their research. They participate in two audio-taped semi-structured interviews that last from about 90 to 120 minutes. They may also participate in one or both of the following optional study components:

* A third semi-structured interview that explores implementing a new method of describing study populations in data analysis.
* 2 to 3 days of lab observation, in which a member of the study research team meets the lab members, observes daily activities and attends lab meetings.

DETAILED DESCRIPTION:
The usefulness of social and political population labels, including those based on race, ethnicity, geographic location, ancestry, and nationality, in science and medicine is a topic of heated debate. The discussion is significant not only for defining rigorous scientific study designs, but for influencing how scientists and the broader society conceptualize, discuss, and react to human difference. Misuse of population descriptors in genetic and genomic research has the potential to perpetuate misinformation, stigmatize certain groups and simplify the complex relationships between individual identity, genetics, and health. With such potential harms in mind, National Institutes of Health guidelines to use the Office of Management and Budget categories of race and ethnicity to monitor inclusion in clinical trials and evaluate potential differences in the safety and efficacy of interventions have been questioned. As increasing attention is given to the implications of human genetic variation on disease and health, actively engaging with scientists may help to identify a lexicon for discussing human genetic variation that is scientifically sound and socially and politically meaningful. We aim to conduct a pilot qualitative study of genetic researchers, exploring their use of population descriptors in human genetic research, including an experiment in which they have the opportunity to describe and group their study populations in a new way. We use qualitative methods to capture researchers' opinions and practices as they think critically about the use of population labels in their studies. Understanding individual scientists opinions about the strengths and weaknesses of different classifications in various contexts will provide important data to help define and facilitate appropriate use of population descriptors in human genetic research.

ELIGIBILITY:
* INCLUSION CRITERIA:

The study population is comprised of intramural and extramural principal investigators:

* Conducting human genetic or genomic research on common disease
* Conducting a project in which they use population descriptors to describe their study sample
* Have collected, at a minimum, preliminary data that allows them to complete an exploratory exercise re-conceptualizing their use of population descriptors in this project.

Participation is limited to researchers who have collected data that gives them sufficient background and context to meaningfully complete this exercise. Insight gathered from our study population on alternatives to existing methods of population classification and description used in human genetic research is especially useful not only because of their professional expertise, but because they are the group that would need to implement alternatives.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-09-18; Study Completion 2012-08-08

CONTACTS AND LOCATIONS:
Overall Officials: Vence L Bonham, J.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pennisi E. Breakthrough of the year. Human genetic variation. Science. 2007 Dec 21;318(5858):1842-3. doi: 10.1126/science.318.5858.1842. PMID 18096770
- [Background] Burchard EG, Ziv E, Coyle N, Gomez SL, Tang H, Karter AJ, Mountain JL, Perez-Stable EJ, Sheppard D, Risch N. The importance of race and ethnic background in biomedical research and clinical practice. N Engl J Med. 2003 Mar 20;348(12):1170-5. doi: 10.1056/NEJMsb025007. No abstract available. PMID 12646676
- [Background] Tang H, Quertermous T, Rodriguez B, Kardia SL, Zhu X, Brown A, Pankow JS, Province MA, Hunt SC, Boerwinkle E, Schork NJ, Risch NJ. Genetic structure, self-identified race/ethnicity, and confounding in case-control association studies. Am J Hum Genet. 2005 Feb;76(2):268-75. doi: 10.1086/427888. Epub 2004 Dec 29. PMID 15625622